CLINICAL TRIAL: NCT06272851
Title: Comparing the Choroidal Thickness Using Optical Coherence Tomography Between the Eyes of Healthy Individuals and Diabetic Patients Without Retinopathy
Brief Title: Measuring Choroidal Thickness Using Optical Coherence Tomography
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nancy Basem Monier, NBMonier, Assiut University
Other Study IDs: Choroidal thickness by OCT
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Choroid Disease; Diabetes Mellitus
MeSH Terms: conditions — Choroid Diseases; Diabetes Mellitus | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diabetics: Type 2 DM patients aged 30 to 80 years
  Interventions: Device: optical coherence tomography
- non diabetics: non-diabetic healthy individuals
  Interventions: Device: optical coherence tomography

INTERVENTIONS:
Device: optical coherence tomography — measuring choroidal thickness using optical coherence tomography

SUMMARY:
To compare the choroidal thickness in eyes of diabetic patients with eyes of age matched controls using optical coherence tomography.

DETAILED DESCRIPTION:
Diabetic retinopathy (DR) is the most common and specific complication of DM. It is one of the leading causes of preventable blindness in the adult working population. (1) DR was the fifth leading cause of blindness and of moderate and severe vision impairment.

Global prevalence of diabetic retinopathy was 22.27% and prevalence was highest in Africa (35.90%). (1)

Fortunately, much of the visual loss from DR is preventable, and the rates of vision loss from diabetes and DR have declined over the past few decades due to advances in ocular disease assessment, screening, imaging and treatment in recent years. (2)

The outer third of the retina gets oxygen and nutrients from choroid. The three vascular layers of choroid are chorio capillaries layer, Sattler layer and Haller layer. (3)

A healthy choroid is essential for retinal function by continuous perfusion into the outer retina, which plays critical roles in thermoregulation of the retina, maintenance of the anatomic position of the retina, removal of residues, and secretion of growth factors. (4-5)

The vascular choroid changes of the diabetic patients are quite similar to those seen in DR, such as increased vascular tortuosity, vascular outpouchings, microaneurysms, nonperfusion areas, vascular dilations and narrowing, and choroidal neovascularization. (6)

Until recently, the choroid could only be evaluated by indocyanine green angiography, laser Doppler flowmetry, and ultrasonography. (6) Optical coherence tomography (OCT) is a non-invasive imaging modality, which is used in acquiring high-resolution sections of retina. (5)

ELIGIBILITY:
Inclusion Criteria:

* All known Type 2 DM patients aged 30 to 95 years either gender who presented to ophthalmology clinics in Assuit ophthalmology hospital with no history of ocular treatment (ocular treatment naïve) and visual acuity of 0.1 (6/60) or more that are able to complete an eye examination, and non-diabetic healthy individuals (HbA1c <7) will be included in the study.

Exclusion Criteria:

* Known diagnosis of any other retinal disease, glaucoma, neurodegenerative disease, and any significant media opacities that precluded fundus imaging and not giving consent will be excluded.

Ages: 30 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: known Type 2 DM patients aged 30 to 95 years either gender with no history of ocular treatment and non-diabetic healthy individuals who come to the hosoital
Sampling Method: Non-Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2029-03-30 (Estimated); Study Completion 2029-05-15 (Estimated)

PRIMARY OUTCOMES:
comparison between choroidal thickness | 2 years
  To compare choroidal thickness using optical coherence tomography between eyes of healthy individuals and diabetic patients without retinopathy

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Shehata Hussein, Study Director — Assiut University; Dalia Mohamed El-Sebaity, Study Director — Assiut University

REFERENCES:
- [Background] Teo ZL, Tham YC, Yu M, Chee ML, Rim TH, Cheung N, Bikbov MM, Wang YX, Tang Y, Lu Y, Wong IY, Ting DSW, Tan GSW, Jonas JB, Sabanayagam C, Wong TY, Cheng CY. Global Prevalence of Diabetic Retinopathy and Projection of Burden through 2045: Systematic Review and Meta-analysis. Ophthalmology. 2021 Nov;128(11):1580-1591. doi: 10.1016/j.ophtha.2021.04.027. Epub 2021 May 1. PMID 33940045
- [Background] Tan TE, Wong TY. Diabetic retinopathy: Looking forward to 2030. Front Endocrinol (Lausanne). 2023 Jan 9;13:1077669. doi: 10.3389/fendo.2022.1077669. eCollection 2022. PMID 36699020
- [Background] Hassan H, Cheema A, Tahir MA, Nawaz HN. Comparison of choroidal thickness in eyes of diabetic patients with eyes of healthy individuals using optical coherence tomography in a tertiary care hospital. Pak J Med Sci. 2022 Jan-Feb;38(1):254-260. doi: 10.12669/pjms.38.1.4443. PMID 35035435
- [Background] Endo H, Kase S, Saito M, Yokoi M, Takahashi M, Ishida S, Kase M. Choroidal Thickness in Diabetic Patients Without Diabetic Retinopathy: A Meta-analysis. Am J Ophthalmol. 2020 Oct;218:68-77. doi: 10.1016/j.ajo.2020.05.036. Epub 2020 Jun 20. PMID 32574782
- [Background] Regatieri CV, Branchini L, Carmody J, Fujimoto JG, Duker JS. Choroidal thickness in patients with diabetic retinopathy analyzed by spectral-domain optical coherence tomography. Retina. 2012 Mar;32(3):563-8. doi: 10.1097/IAE.0b013e31822f5678. PMID 22374157
- [Background] Tavares Ferreira J, Vicente A, Proenca R, Santos BO, Cunha JP, Alves M, Papoila AL, Abegao Pinto L. CHOROIDAL THICKNESS IN DIABETIC PATIENTS WITHOUT DIABETIC RETINOPATHY. Retina. 2018 Apr;38(4):795-804. doi: 10.1097/IAE.0000000000001582. PMID 28267113